CLINICAL TRIAL: NCT01655147
Title: An Open-Label Drug-Drug Interaction Study to Assess the Effect of Rifampicin on the Pharmacokinetics of Abiraterone (JNJ-589485) Following Administration of Abiraterone Acetate (JNJ-212082) Tablets in Healthy Male Subjects
Brief Title: A Study to Evaluate the Effect of Rifampicin on the Pharmacokinetics of Abiraterone in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100651; 212082PCR1003 (Other: Janssen Research & Development, LLC); 2011-003490-28 (EudraCT Number)
Record Dates: First submitted 2012-01-23; First posted 2012-08-01 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Healthy; Pharmacokinetics; Abiraterone acetate; Abiraterone; JNJ-589485; JNJ-212082; Zytiga; Rifampicin; Rifadin; CYP3A4 inducer
MeSH Terms: interventions — Abiraterone Acetate; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate + Rifampicin (Experimental): Abiraterone acetate 1,000 mg (4 x 250 mg) on Day 1 of Period 1. Rifampicin 600 mg (2 x 300 mg) on Days 8 to 13, and Abiraterone acetate 1,000 mg (4 x 250 mg) on Day 14 of Period 2.
  Interventions: Drug: Abiraterone acetate; Drug: Rifampicin

INTERVENTIONS:
Drug: Abiraterone acetate — Type=exact number, unit=mg, number=1,000, form=tablet, route=oral. Abiraterone acetate administered on Day 1 of Period 1, and Day 14 of Period 2.
  Other Names: ZYTIGA
Drug: Rifampicin — Type=exact number, unit=mg, number=600, form=capsule, route=oral. Rifampicin administered on Days 8 to 13 of Period 2.
  Other Names: RIFADIN

SUMMARY:
The purpose of this study is to assess the effects of repeated daily administration of rifampicin on the pharmacokinetics (what the body does to the medication) of abiraterone following single-dose administration of abiraterone acetate tablets in healthy male participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center (study conducted at one site), 2-period, sequential-design (studies that combine both longitudinal and cross sectional methods), to evaluate the effects of rifampicin on the pharmacokinetics of abiraterone acetate in healthy male participants. The study consists of a screening phase, an open-label treatment phase, and a follow up phase. The screening phase will be within 14 days before the first study medication administration. The treatment phase will consist of 2 treatment periods, Period 1: a single oral dose of abiraterone acetate tablets, and Period 2: a daily oral dose of rifampicin capsules alongwith a single oral dose of abiraterone acetate tablets. The 2 periods will be separated by a washout period of at least 7 days. Blood sample collection for pharmacokinetic assessments will be done for determination of abiraterone and rifampicin concentrations. The follow up phase will be of 14 days. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examinations will be monitored throughout the study. The total study duration will be approximately 31 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* Must have a 12-lead electrocardiogram consistent with normal cardiac conduction and function
* Must sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Must agree to use an adequate contraception method and to not donate sperm during the study and for 3 months after receiving the last dose of study medication
* Have willingness to participate in the optional pharmacogenomic component of this study, participants (or their legally acceptable representative) must have signed the informed consent form

Exclusion Criteria:

* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, and others
* Clinically significant abnormal values for hematology or clinical chemistry at screening or at admission to the study center
* Serum testosterone level of < 200 ng/dL (at screening)
* Clinically significant renal laboratory findings including specifically, creatinine, and creatinine clearance
* Clinically significant hepatic laboratory findings or signs

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of abiraterone in Period 1 and Period 2 | Period 1: Day 1 to Day 4; Period 2: Day 14 to Day 17
  Pharmacokinetic parameter Cmax of abiraterone was measured when abiraterone acetate was administered in Period 1 and Period 2.
Area under the plasma concentration-time curve (AUC) of abiraterone in Period 1 and Period 2 | Period 1: Day 1 to Day 4; Period 2: Day 14 to Day 17
  Pharmacokinetic parameter AUC of abiraterone was measured when abiraterone acetate was administered in Period 1 and Period 2.
Time to reach the maximum plasma concentration (tmax) of abiraterone in Period 1 and Period 2 | Period 1: Day 1 to Day 4; Period 2: Day 14 to Day 17
  Pharmacokinetic parameter tmax of abiraterone was measured when abiraterone acetate was administered in Period 1 and Period 2.
Eliminaton half-life (t1/2) of abiraterone in Period 1 and Period 2 | Period 1: Day 1 to Day 4; Period 2: Day 14 to Day 17
  Pharmacokinetic parameter t1/2 of abiraterone was measured when abiraterone acetate was administered in Period 1 and Period 2.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium